CLINICAL TRIAL: NCT03938077
Title: A Community-University Approach to Preventing HIV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unfortunately, the co-PI and lead community partner relocated out of the target area. Therefore, recruiting participants from the target area was not feasible.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, David Cordova, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00151011
Record Dates: First submitted 2019-04-15; First posted 2019-05-06 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: HIV/AIDS and Infections; Drug Abuse; Adolescent Behavior; Drug Usage; Alcohol Use; Mental Health; Tobacco Use; HIV Testing
Keywords: mHealth; prevention intervention; primary health care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections; Substance-Related Disorders; Adolescent Behavior; Alcohol Drinking; Psychological Well-Being; Tobacco Use

STUDY DESIGN:
Intervention Model Description: To examine the preliminary efficacy of the S4E intervention in improving the uptake of HIV self-testing immediately post-intervention and the feasibility(e.g., enrollment rates, eligibility) and acceptability (e.g., satisfaction) of S4E .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- S4E App intervention (Experimental): Youth will receive the S4E intervention via provided iPads. The intervention will last approximately 60. Content includes: (a) storytelling scenarios, (b) drug use and HIV/STI knowledge, (c) interactive activities, (d) increasing self-efficacy to prevent/reduce sexual and drug use risk behaviors and increase HIV self-testing, (e) Near Peer-youth communication, and (f) highlighting prevention principles. The youth will participate in a Near Peer-initiated prevention and risk reduction encounter which includes (a) reinforcement of HIV solutions that youth learned in the S4E app, (b) promotion of HIV self-tests, and (c) linkage to care and prevention services.
  Youth have the option to take a HIV self-test. We will determine the acceptability of youth disclosing their results to their Near Peer and linkage to resources.
  The research staff will also conduct in-depth qualitative interviews with both youth and Near Peer participants to assess feasibility and acceptability of S4E.
  Interventions: Device: Storytelling 4 Empowerment

INTERVENTIONS:
Device: Storytelling 4 Empowerment — S4E application was developed in collaboration with youth in Southeast Michigan. S4E aims to prevent and reduce HIV/STI risk behaviors, including drug use and sexual risk behaviors, and increase HIV testing among youth. Content produced for the application is based on scientific prevention principles in conjunction with youth input. To date, we have developed modules focused on youth alcohol & drug use, HIV & STIs, and tobacco prevention and cessation.

SUMMARY:
Examine the feasibility and acceptability of delivering the S4E intervention to 20 African-American youths between the ages 16-21 in Flint, Michigan. The investigators will examine the preliminary efficacy of the S4E intervention in improving the uptake of HIV self-testing immediately post-intervention.

DETAILED DESCRIPTION:
HIV is a significant public health concern in the US, and African American youth (defined as the adolescent and young adults 16-21 years of age) are disproportionately affected. Furthermore, HIV risk behaviors, including substance use and sexual risk behaviors are prominent. Despite the disproportionately high rates of HIV infection and risk behaviors in youth, few youth report having ever been tested for HIV and many are not routinely screened for asymptomatic STIs as recommended by the Center for Disease Control. To address these significant public health concerns, a mobile-health (mHealth) intervention, Storytelling 4 Empowerment (S4E) was developed for health clinic settings. S4E has demonstrated high feasibility, acceptability, and preliminary efficacy among youth in clinic settings. The proposed research will determine the feasibility and acceptability of delivering S4E via near peers, as well as determine the preliminary efficacy of S4E to improve HIV self-testing immediately post-intervention in a community sample (n=20) of at-risk youth ages 16-21 living in Flint, Michigan by conducting a phase I, one-arm pilot study to examine the feasibility and preliminary efficacy of S4E in improving the uptake of HIV self-testing immediately post-intervention. A University-Community approach was taken to employ principles of Community Based Participatory Research (CBPR) to determine the accessibility and acceptability of S4E when delivered by Near Peers.

ELIGIBILITY:
Inclusion Criteria:

* 16-21 years of age
* Sexually Active
* African American
* Live in Flint Michigan

Exclusion Criteria:

* Report of prior psychiatric hospitalization by adolescent
* Visible cognitive impairment due to drug use

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Lifetime HIV Testing | Baseline
  At baseline we will assess binary outcome of participant's lifetime HIV testing and collect date of most recent HIV test using an item adapted from the Centers for Disease Control (CDC) Youth Behavior Risk Survey (YRBS). A sample question for youth is "Have you every been tested for HIV?". Responses consist of "1=Yes", "0=No", and "98=Refuse to Answer".
HIV Self-Testing | Immediately post-intervention
  Immediately post-intervention, we will assess the binary outcome of HIV self-testing using items adopted from Lightfoot and colleagues (2018).
HIV Self-Test Results Disclosure | Immediately post-intervention
  Post-intervention we will asses the percentage of youth that disclose their HIV self-test results to the Near Peer.

SECONDARY OUTCOMES:
Change in Sexual Risk Beliefs from baseline to immediately post-intervention | baseline and immediatly post-intervention
  Beliefs regarding sexual behaviors (e.g., intended sex, condom use, and other contraceptives) will be assessed. A sample question for the youth is, "Condoms help prevent pregnancy." Responses range from "1=Strongly disagree" to "5=Strongly Agree".
Change in Sexual Risk Attitudes from baseline to immediately post-intervention | baseline and immediatly post-intervention
  Attitudes about sexual behaviors (e.g., intended sex, condom use, and other contraceptives) will be assessed. A sample question for the youth is "If I used a condom, sex would not feel as good." Responses range from "1=Strongly disagree" to "5=Strongly Agree".
Change in Future intentions regarding sexual risk from baseline to immediately post-intervention | baseline and immediatly post-intervention
  Change in future intentions of sexual behaviors (e.g., intended sex, condom use, and other contraceptives) will be assessed. A sample question for the youth is, "How likely is it that you will decide to have sex in the next 90 days?"." Responses range from "1=Very Unlikely" to "5=Very Likely".
Linkage to Care and Prevention | immediately post-intervention
  The percent of youth who are referred to substance use, mental health, and sexual health services will be assessed.
Eligibility rates for the Near Peer | enrollment period pre-intervention
  During the recruitment period of Near Peers, we will monitor and record the percentage of potential near peer participants who meet eligibility criteria to be enrolled in the study.
Percent of Enrollment for Near Peer | enrollment period pre-intervention
  During the recruitment period of Near Peers, we will monitor and record the percentage of those potential near peers eligible to participate who decide to enroll in the study.
Intervention Completion Rates for Near Peer | immediately-post intervention
  Immediately post intervention we will assess the rate of intervention completion of Near Peers.
Eligibility rates for the Youth | enrollment period pre-intervention
  Immediately post-intervention, we will assess the percentage of participants who meet eligibility criteria for our study.
Percent of Enrollment for Youth | enrollment period pre-intervention
  We will assess the percentage of those youth eligible to participate who are enrolled in the study.
Intervention Completion Rates for Youth | immediately post-intervention
  Immediately post intervention, we will assess the rate of intervention completion of youth participants.
Near Peer Satisfaction of the S4E app: Client Satisfaction Questionnaire (CSQ) | immediately-post intervention
  Satisfaction is defined as how much the Near Peer enjoyed using the app and will be measured by the Client Satisfaction Questionnaire (CSQ). The CSQ is a eight item survey adapted from Larsen and colleagues (1979) that has been shown to be reliable and valid, and was previously used in a primary care intervention (Cordova et al., 2018). In our previous studies the alphas have ranged from 0.87 to 0.92. A sample question is "How would you rate the app you have received?". Responses range from "1=Poor" to "4=Excellent".
Acceptability of S4E Session for Near Peer: Session Evaluation Form (SEF) | immediately-post intervention
  Acceptability is defined as how much the Near Peer enjoyed the intervention and will be measured by the Session Evaluation Form (SEF). The SEF is a 13-item survey, modified from Harper and colleagues (2008), that has been shown to be reliable and valid, and was previously used in a primary care intervention (Cordova et al., 2018). In our previous studies the alpha of SEF was 0.89. A sample question is "The session was enjoyable". Responses range from "1=Strongly Agree" to "4=Strongly Disagree".
Youth Satisfaction of the S4E app: Client Satisfaction Questionnaire (CSQ | immediately-post intervention
  Satisfaction is defined as how much the youth enjoyed using the app and will be measured by the Client Satisfaction Questionnaire (CSQ). The CSQ is a eight item survey adapted from Larsen and colleagues (1979) that has been shown to be reliable and valid, and was previously used in a primary care intervention (Cordova et al., 2018). In our previous studies the alphas have ranged from 0.87 to 0.92. A sample question is "How would you rate the app you have received?". Responses range from "1=Poor" to "4=Excellent".
Acceptability of S4E Session for Youth: Session Evaluation Form (SEF) | immediately-post intervention
  Acceptability is defined as how much the youth enjoyed the interview session and will be measured by the Session Evaluation Form (SEF). The SEF is a 13-item survey, modified from Harper and colleagues (2008), that has been shown to be reliable and valid, and was previously used in a primary care intervention (Cordova et al., 2018). In our previous studies the alpha of SEF was 0.89. A sample question is "The session was enjoyable". Responses Range from "1=Strongly Agree" to "4=Strongly Disagree".

OTHER OUTCOMES:
Change in Near Peer-Youth Communication for Near Peers from baseline to immediately post-intervention | baseline and immediately post-intervention
  Completed by the Near Peer, Near Peer-youth communication will be assessed post-baseline using items adapted from the Matched Pair Instrument (19 items; MPI). MPI assesses process and content of communication, including verbal and action-related behaviors performed by Near Peers. Responses range from "1=strongly disagree," to "5=strongly agree," on a five-point Likert scale. A sample statement for Near Peers and youths is, " I encouraged the youth to express his or her thoughts concerning drug use behaviors."
  The Adolescent Patient-Provider Interaction Scale will also be used to assess Near Peer- youth interaction for accessing sexual and reproductive health care (e.g., the Near Peer explained everything youth needed to know).
Change in Near Peer-Youth Communication for Youth from baseline to immediately post-intervention | baseline and immediately post-intervention
  Completed by the youth, Near Peer-youth communication will be assessed post-baseline using items adapted from the Matched Pair Instrument (19 items; MPI). MPI assesses process and content of communication, including verbal and action-related behaviors performed by Near Peers. Responses range from "1=strongly disagree," to "5=strongly agree," on a five-point Likert scale. A sample statement for Near Peers and youths is, "I was encouraged to express my thoughts concerning drug use behaviors."
  The Adolescent Patient-Provider Interaction Scale will also be used to assess Near Peer- youth interaction for accessing sexual and reproductive health care (e.g., the Near Peer explained everything youth needed to know).
Change in Youth Self-Efficacy as measured by Drug Use Resistance Self-Efficacy Scale from baseline to immediately post-intervention | baseline and immediately post-intervention
  Youth's self-efficacy will be assessed using two scales, including the Condom Self-Efficacy Scale (19 items, α =.85), and Drug Use Resistance Self-Efficacy (24 items, α =.98). Responses range from "1=not sure at all," to "4=definitely sure," on a four-point Likert scale. A sample question for the youth is, "How sure are you that you can refuse if a friend offers you marijuana at a party and you do not want it?"
Change in Youth Self-Efficacy as measured by the Condom Self-Efficacy Scale from baseline to immediately post-intervention | baseline and immediately post-intervention
  Youth's self-efficacy will be assessed using two scales, including the Condom Self-Efficacy Scale (19 items, α =.85), and Drug Use Resistance Self-Efficacy (24 items, α =.98). Responses range from "1=not sure at all," to "4=definitely sure," on a four-point Likert scale. A sample question for the youth is, "How sure are you that you can refuse if a friend offers you marijuana at a party and you do not want it?"

CONTACTS AND LOCATIONS:
Overall Officials: David Cordova, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - YOUR Center, Flint, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cordova D, Alers-Rojas F, Lua FM, Bauermeister J, Nurenberg R, Ovadje L, Fessler K, Delva J, Salas-Wright CP, Council YL. The Usability and Acceptability of an Adolescent mHealth HIV/STI and Drug Abuse Preventive Intervention in Primary Care. Behav Med. 2018 Jan-Mar;44(1):36-47. doi: 10.1080/08964289.2016.1189396. Epub 2016 Jul 15. PMID 27223646
- [Background] Cordova D, Bauermeister JA, Fessler K, Delva J, Nelson A, Nurenberg R, Mendoza Lua F, Alers-Rojas F, Salas-Wright CP; Youth Leadership Council. A Community-Engaged Approach to Developing an mHealth HIV/STI and Drug Abuse Preventive Intervention for Primary Care: A Qualitative Study. JMIR Mhealth Uhealth. 2015 Dec 18;3(4):e106. doi: 10.2196/mhealth.4620. PMID 26685288
- [Background] Cordova D, Lua FM, Ovadje L, Fessler K, Bauermeister JA, Salas-Wright CP, Vaughn MG, Leadership Council Y. Adolescent Experiences of Clinician-Patient HIV/STI Communication in Primary Care. Health Commun. 2018 Sep;33(9):1177-1183. doi: 10.1080/10410236.2017.1339379. Epub 2017 Jul 7. PMID 28686489